CLINICAL TRIAL: NCT05587478
Title: A Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled, First-In- Human Study of Orally Administered EDP-323 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses, Multiple Ascending Doses, and the Effect of Food on EDP-323 Pharmacokinetics in Healthy Participants
Brief Title: A Study of EDP-323 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDP 323-001
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-10

CONDITIONS: RSV Infection
Keywords: First-in-Human; Single Ascending Dose; Multiple Ascending Dose; Healthy Volunteer
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- EDP-323 SAD Cohorts (Experimental): EDP-323 Dose 1, Dose 2, Dose 3, Dose 4, Dose 5 and Dose 6, orally, once daily in one single administration
  Interventions: Drug: EDP-323
- EDP-323 MAD Cohorts (Experimental): EDP-323 Dose 1, Dose 2, Dose 3 and Dose 4 orally, once daily for 7 days
  Interventions: Drug: EDP-323
- EDP-323 SAD Placebo Cohorts (Placebo Comparator): Matching placebo, orally, once daily in one single administration
  Interventions: Drug: Placebo
- EDP-323 MAD Placebo Cohorts (Placebo Comparator): Matching placebo, orally, once daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-323 — Oral administration
  Arms: EDP-323 MAD Cohorts; EDP-323 SAD Cohorts
Drug: Placebo — Placebo to match EDP-323, oral administration
  Arms: EDP-323 MAD Placebo Cohorts; EDP-323 SAD Placebo Cohorts

SUMMARY:
This study is a randomized, double-blind, sponsor-open, placebo-controlled study. It will assess the safety, tolerability, and pharmacokinetics of orally administered single and multiple doses of EDP-323 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 65 years, inclusive.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* Infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) at screening and infection with SARS-CoV-2 at the Day -1 visit
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Receipt of any vaccine, an investigational agent or biological product within 28 days or 5 times the t½, whichever one is longer, prior to first dose.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Safety measured by adverse events | Up to 8 Days in SAD Cohorts
Safety measured by adverse events | Up to 14 Days in MAD Cohorts

SECONDARY OUTCOMES:
Cmax of EDP-323 | Up to 5 Days in SAD Cohorts
AUC of EDP-323 | Up to 5 Days in SAD Cohorts
Cmax of EDP-323 | Up to 11 Days in MAD Cohorts
AUC of EDP-323 | Up to 11 Days in MAD Cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- ICON, plc., Lenexa, Kansas, United States